CLINICAL TRIAL: NCT05028179
Title: PROTEUS: A PROspective Randomised Controlled Trial Evaluating the Use of Artificial Intelligence in Stress Echocardiology
Brief Title: PROTEUS: Evaluating the Use of Artificial Intelligence to Support Stress Echocardiography Testing for Heart Disease
Acronym: PROTEUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ultromics Ltd (Industry)
Collaborators: University of Oxford (Other); Academic Health Science Centres (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: COL-69
Record Dates: First submitted 2021-07-22; First posted 2021-08-31 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: A multi-centre, two-arm, randomised controlled trial. Randomised 1:1
  * Standard care group (comparator)
  * Standard care plus AI platform (EchoGo)
Who Masked: Participant
Masking Description: Following the stress echocardiogram examination, participants will follow the care pathway determined by the clinical team managing their care. If the participant is assigned to the study intervention arm the EchoGo report will inform this decision making process.
  In order to minimise bias in any outcome assessment clinicians will be asked not to share the details of the EchoGo report received for participants within the intervention arm with the participant or with colleagues who may undertake future investigations eg: angiography.If a clinician subsequently considers there is a clinical need to know the details of the EchoGo report this can be made available at the discretion of the study team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (comparator) (No Intervention): Patients will receive standard care
- Standard Care plus AI platform (EchoGo) (Experimental): Patients will receive standard care plus their Echocardiogram will be sent to Ultromics for AI assessment. The report from the assessment will be sent to the clinician, and utilised to inform the patients further care.
  Interventions: Diagnostic Test: EchoGo

INTERVENTIONS:
Diagnostic Test: EchoGo — EchoGo Pro is an software Medical Device which is able to assess Stress Echocardiograms and provide a binary classification of risk of CAD
  Arms: Standard Care plus AI platform (EchoGo)

SUMMARY:
PROTEUS is a multicentre, two arm, randomised controlled trial of a medical device to assess the impact of the introduction of EchoGo into the standard care pathway for stress echocardiology.

DETAILED DESCRIPTION:
Title: A Prospective Randomised Controlled Trial Evaluating the Use of AI in Stress Echocardiography

Trial design: Multi-centre, two-arm, Randomised Controlled Trial of a medical device. Randomised 1:1 to either:

* Standard care (comparator), or
* Standard care plus AI Platform (EchoGo) Trial participants: Adults undergoing clinically indicated stress echocardiogram (SE) to assess inducible ischaemia at participating NHS Trusts.

Having benchmarked the device performance (Upton 2019), and having successfully deployed and tested the required infrastructure, we now propose to prospectively test the software in clinical practice. Based on the existing data for accuracy we would expect use of the EchoGo Platform in the clinical pathway will have a significant benefit reducing inter-reader variability, increasing accuracy and thereby reducing health costs. To formally evaluate the impact of automated AI quantification and accuracy of the decision to make a referral to coronary angiogram, following stress echocardiography, we propose a prospective, multi-centre, randomised controlled trial that compares provision of an AI derived report to a clinician against clinician-only standard of care. This will provide the highest level of evidence of any potential benefit or disadvantages prior to adoption of the software for widespread clinical implementation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Male or female, ≥18 years of age at study entry
* Referred to an NHS Trust for stress echocardiography for investigation of ischaemic heart disease

Exclusion Criteria:

* More than moderate valvular heart disease
* Left ventricular outflow tract obstruction defined as a gradient > 30mmHg (fixed or dynamic; supravalvular, valvular or sub-valvular)
* Significant co-morbidities (e.g. cancer) with an expected life-expectancy of under 12 months in the investigator's opinion
* Previous coronary artery bypass graft or other cardiac surgery
* Congenital or inherited myocardial disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2338 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Investigate if EchoGo plus standard care is non-inferior to standard care alone for aiding referral to coronary angiogram following stress echocardiogram (SE) | 6 months post stress echo
  Outcome measure - AUROC for the ability to make an appropriate referral to coronary angiogram at 6 months following stress echocardiogram.
  Appropriate management will be defined as a composite of
  * coronary angiography that demonstrates severe coronary disease fulfilling clinical care guidelines for revascularisation or
  * decision for medical management/reassurance without unanticipated serious adverse cardiac events Outcome data will be collected from participant's medical records at 3 and 6 months.

SECONDARY OUTCOMES:
Investigate if EchoGo plus standard care is superior to standard care alone in predicting the risk of severe cardiovascular disease following stress echocardiogram (SE) | 6 month post stress echo
  Outcome shall be measured through - AUROC for the ability to make an appropriate referral to coronary angiogram.
Investigate the appropriate clinical management decisions made when using EchoGo plus standard care compared to standard care alone. | 6 month post stress echo
  Outcome measure - Appropriate clinical management following an echocardiogram, for referring a patient to coronary angiogram, determined by adjudication committee review of follow up data.
Establish if clinical management decision making is affected by review of the EchoGo report. | 6 month
  Establish if clinical management decision making is affected by review of the EchoGo report as recorded by clinician self-report.
Establish if using the EchoGo platform affects clinician diagnostic confidence. | 3 and 6 months post stress echo
  Clinician diagnostic confidence in their interpretation of the stress echo report will be measured by clinician self-report at baseline, 3 months and end of study at each participating site.
Establish if clinician diagnostic performance variance reduces with EchoGo use. | 3 and 6 month post stress echo
  Outcome measured by Inter-clinician and in-site variability at baseline, 3 months and at end of study.
Establish if using Ultromics' EchoGo Platform affects the number of subsequent investigations for cardiovascular disease. for cardiovascular disease | 3 and 6 months post stress echo
  Outcome shall be measured through collation of the number of incidences of the following (occurring up to 6 months following stress echo):
  * Myocardial Perfusion Scan
  * CT coronary angiogram
  * Stress echo
  * Invasive coronary angiogram
  * Stress CMR
  * Exercise tolerance test
  * Initiation of anti-anginal medication/medical management of angina
  Data will be collected from participants medical records at 3 and 6 months
Establish if using Ultromics' EchoGo Platform affects patient reported coronary artery disease symptoms. | 3 and 6 months post stress echo
  Outcome shall be measured through the collation of the number of coronary artery disease symptoms and impact on participant health status as measured by patient-reported short Seattle Angina Questionnaire (SAQ-7) at trial entry, 3 months and 6 months
Assess the health economics impact of implementation and use of Ultromics' EchoGo platform in NHS units | 3 and 6 month post stress echo
  Outcome measure - Patient reported health related quality of life

CONTACTS AND LOCATIONS:
Locations (20):
- United Kingdom (20):
  - Great Western Hospitals NHS Foundation Trust, Swindon, Oxfordshire
  - Mid and South Essex NHS Foundation Trust, Basildon
  - Royal United Hospitals Bath, Bath
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - University Hospitals Coventry & Warwickshire, Coventry
  - Northumbria Healthcare NHS Foundation Trust, Hexham
  - Buckinghamshire Healthcare NHS Trust, High Wycombe
  - Ipswich General Hospital, Ipswich
  - Leicester General Hospital, Leicester
  - St George's University Hospitals NHS Foundation Trust, London
  - Milton Keynes University Hospital, Milton Keynes
  - Northampton General Hospital NHS Trust, Northampton
  - Royal Oldham Hospital, Oldham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - North West Anglia NHS Foundation Trust, Peterborough
  - Royal Berkshire Hospital, Reading
  - Salford Royal Hospital, Salford
  - Stockport NHS Foundation Trust, Stockport
  - Wrightington, Wigan and Leigh Teaching Hospitals NHS Foundation Trust, Wigan

REFERENCES:
- [Derived] Fazakarley CA, Breen M, Leeson P, Thompson B, Williamson V. Experiences of using artificial intelligence in healthcare: a qualitative study of UK clinician and key stakeholder perspectives. BMJ Open. 2023 Dec 11;13(12):e076950. doi: 10.1136/bmjopen-2023-076950. PMID 38081671
- [Derived] Woodward G, Bajre M, Bhattacharyya S, Breen M, Chiocchia V, Dawes H, Dehbi HM, Descamps T, Frangou E, Fazakarley CA, Harris V, Hawkes W, Hewer O, Johnson CL, Krasner S, Laidlaw L, Lau J, Marwick T, Petersen SE, Piotrowska H, Ridgeway G, Ripley DP, Sanderson E, Savage N, Sarwar R, Tetlow L, Thompson B, Thulborn S, Williamson V, Woodward W, Upton R, Leeson P. PROTEUS Study: A Prospective Randomized Controlled Trial Evaluating the Use of Artificial Intelligence in Stress Echocardiography. Am Heart J. 2023 Sep;263:123-132. doi: 10.1016/j.ahj.2023.05.003. Epub 2023 May 14. PMID 37192698